CLINICAL TRIAL: NCT05880901
Title: Increasing Low-income Children's Access to Healthy Structured Programming to Reduce Obesity
Brief Title: Healthy Kids Beyond the Bell: Investigating the Impact of After-School and Summer Programs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, R. Glenn Weaver, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00125471
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Health Status Disparities; Pediatric Obesity; Ethnic Group; Socioeconomic Factors
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): does not attend afterschool or summer programing
- After school (Experimental): Attends after school programming for 32 weeks during the school year
  Interventions: Behavioral: After school program
- Summer camp (Experimental): Attends summer day camp programming for 8 weeks during the summer vacation from school
  Interventions: Behavioral: Summer day camp
- After school and Summer Camp (Experimental): Attends after school programming for 32 weeks during the school year and summer day camp programming for 8 weeks during the summer vacation from school
  Interventions: Behavioral: After school program; Behavioral: Summer day camp

INTERVENTIONS:
Behavioral: After school program — The after school program are existing community-based programs that take place immediately after the regular school day (typically 3:00-6:00pm); are located in a school; are available daily throughout the academic year (Monday through Friday); and provide a combination of scheduled activities, which include a snack, homework assistance/tutoring, enrichment activities (e.g., arts and crafts, music), and opportunities for children to be physically active.
  Arms: After school; After school and Summer Camp
Behavioral: Summer day camp — The summer day camp programs are existing camps which take place at schools from which children will be recruited. The camps are not singularly focused, such as sport camps or academic only camps. Rather, the camps provide indoor and outdoor opportunities for children to be physically active each day, provide enrichment and academic programming, as well as provide breakfast, lunch, and snacks.
  Arms: After school and Summer Camp; Summer camp

SUMMARY:
Nearly one in five children are obese, and disparities in overweight and obesity between children from low- and middle-to-high-income households persist despite a multitude of school-based interventions. The structured days hypothesis posits that structure within a school day plays a protective role for children against obesogenic behaviors, and, ultimately, prevents the occurrence of excessive weight gain, thus, past school-based efforts are misplaced. This study will provide access to healthy structured programming via vouchers to afterschool programs and summer day camps during two "windows of vulnerability" (ie afterschool and summer) for low-income children.

DETAILED DESCRIPTION:
Despite the public health field's best efforts, disparities in overweight and obesity (OWOB) prevalence between children (6-11) from low- and middle-to-high-income families persist. Previous interventions to address disparate rates of childhood OWOB have focused almost exclusively on school settings. Given that disparities in OWOB persist, current school-based efforts may be misplaced because children engage in more unhealthy behaviors outside of school (e.g., afterschool during weekdays and during the summer). The structured days hypothesis posits that a structure within a day, defined as a pre-planned, segmented, and adult-supervised compulsory environment (like a school day), plays a protective role for children against obesogenic behaviors, and, ultimately, prevents the occurrence of negative health-outcomes, such as, excessive weight gain. Essentially, the structured days hypothesis draws upon concepts in the 'filled-time perspective' literature which posits that time filled with favorable activities cannot be filled with unfavorable activities. There are at least two "windows of vulnerability" for children outside of the school day. These critically important windows include the hours immediately following school (i.e., 3-6pm school days) and the 10 weeks of summer vacation. Programs that can provide a healthy structured environment and prevent unhealthy weight gains exist for both of these time periods (i.e., afterschool programs and summer day camps). Unfortunately, these programs are too expensive for children from low-income families to attend. Thus, this study will rigorously test the impact of providing access to existing, community-operated afterschool and summer programs on weight status (i.e., BMI z-score) and obesogenic behaviors (i.e., physical activity, screen use, diet, and sleep) of elementary children from low-income households. The study will employ a 2x2 full factorial design. The two factors will be access, through vouchers, to structured programming. The four groups will be a no treatment control, afterschool program voucher only, summer day camp voucher only, and vouchers for afterschool and summer day camp combined. The study will accomplish the following specific aims: AIM 1 (Primary): Compare changes in z-BMI among children in the no treatment control, afterschool only, summer camp only, and afterschool and summer day camp combined groups. AIM 2 (Secondary): Compare differences in obesogenic behaviors during the school year and the summer among children in the no treatment control, school only, summer camp only, and afterschool and summer day camp combined intervention groups. AIM 3 (Secondary): Evaluate the cost-effectiveness of delivering the afterschool only, summer camp only, and combined interventions. This study is significant because nearly one in five children are obese, and disparities in OWOB between children from low- and middle-to-high-income households persist despite past school-based interventions. This study is innovative because it represents one of the first attempts to provide access to healthy structured programming during two "windows of vulnerability" for children outside of the school day. Should the proposed intervention strategy prove effective it has the potential to mitigate disparities in OWOB prevalence.

ELIGIBILITY:
Inclusion Criteria:

* k-4th grader in a partner school
* eligible for free and reduced price lunch (a widely recognized indicator of
* socioeconomic level and poverty status)
* parent that indicates "yes' on an informed consent document for participation in the study

Exclusion Criteria:

* Diagnosis of an intellectual disability, such as Down Syndrome, Fragile X, Fetal Alcohol
* a physical disability, such as wheelchair use, that prevents the ability to ambulate without assistance.
* Families who plan to enroll their children in a summer camp or after school program or relocate (i.e., move) during the 14-month period that they participate

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index | End of school year (0 months, start of summer), beginning of school year (3 months, end of summer) and end of following school year (12 months)
  BMI translated into BMI z-scores based on Centers for Disease Control age-sex-specific zBMI growth charts

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weaver RG, Beets MW, Adams EL, Kaczynski AT, Chen B, Armstrong B, Burkart S, Kiely K, Cepni AB, White JW 3rd, Finnegan O, Savidge M, Parker H, Randolph GAT. Rationale and design of Healthy Kids Beyond the Bell: a 2x2 full factorial study evaluating the impact of summer and after-school programming on children's body mass index and health behaviors. Trials. 2024 Oct 24;25(1):714. doi: 10.1186/s13063-024-08555-2. PMID 39449089